CLINICAL TRIAL: NCT07255924
Title: Anesthesia, Perfusion, and Surgical practicEs in Cardiac Surgery: an Adaptive, Prospective, International, Multicenter, Observational Study.
Brief Title: Anesthesia, Perfusion, and Surgical practicEs in Cardiac Surgery
Acronym: APECx
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Amsterdam UMC, location AMC (Other); VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Nimrat Grewal, Professor and Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2025.0597
Record Dates: First submitted 2025-11-14; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Anaesthesia; Cardiac Surgery; Perfusion; Anesthesia
Keywords: Cardiac Surgery; Cardiac Anaesthesia; Anesthesia; Perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Phase 1: The Phase 1 cohort comprises all participants enrolled during the first phase of the APECx study. The primary focus for this phase/group is to identify global mechanical ventilation strategies and their associations with key clinical outcomes, including the incidence of post-operative pulmonary complications.

SUMMARY:
Perioperative management in cardiac surgery, particularly the use of anesthesia, cardiopulmonary bypass (CPB), and surgical techniques, remains highly variable across institutions. Current international guidelines lack clear recommendations due to insufficient high-quality comparative data. APECx is an adaptive, international, multicenter, prospective, observational study designed to address multiple of these evidence gaps. The adaptive design allows the study to proceed through subsequent phases. Each phase will collect comprehensive global data on specific peri-operative practices and their associated patient outcomes, all within a single, continuously evolving study.

DETAILED DESCRIPTION:
The perioperative management, particularly the use of anesthesia, cardiopulmonary bypass (CPB) and surgical techniques in cardiac surgery, remains highly variable across institutions and regions. Current international guidelines lack clear recommendations due to the insufficiency of high-quality comparative data. Furthermore, over two thirds of the recommendations continue to rely on expert opinion, with little change over time. Given the complexity and physiological burden of cardiac surgery, understanding global variation in anesthetic, perfusion and surgical strategies is critical.

The APECx initiative is an adaptive, international, multicenter, prospective cohort study designed to address multiple of these knowledge gaps. The study aims to promote consistent, evidence-based care by describing global practice variationsand identifying potential modifiable factors that are associated with clinical outcomes.

The core feature of the APECx study is its adaptive design that allows the research focus to evolve over time. The study will proceed through distinct phases, beginning in 2026. Each phase will span approximately one year, concluding once the phase-specific, predefined sample size is reached, at which point the study will transition to the next phase. This framework enables the collection of comprehensive data on specific practices and outcomes within a single, continuously evolving study. To ensure transparency and reproducibility, a detailed protocol for each study phase will be registered on ClinicalTrials.gov prior to phase start.

All data will be prospectively collected by local investigators and entered into a web-based electronic Case Report Form (eCRF) using Castor (Castor Electronic Data Capture, Amsterdam, the Netherlands). Data collection will occur biannually, with participating centers collecting data for a period of two consecutive weeks within a designated three-month window. Follow-up will continue for 30 days post-surgery or until hospital discharge, whichever comes first.

This study will be conducted at cardiac surgery centers worldwide. An inclusive enrollment strategy aims to recruit a broad spectrum of centers, varying in research involvement, surgical complexity, annual caseload, and geographic location, to ensure a globally representative dataset. Centers will have the flexibility to join or leave the study at the beginning of each new phase, a design feature intended to lower the threshold for participation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing cardiac surgery at a participating center

Exclusion Criteria:

- Transcatheter cardiac interventions or endovascular procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing cardiac surgery at one of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | From date of cardiac surgery until hospital discharge, assessed up to 30 days postoperatively.
  Hospital length of stay (LOS) refers to the total duration (in days) of a patient's admission in the hospital.
Intensive Care Unit (ICU) length of stay | From the time of ICU admission immediately after cardiac surgery until transfer out of the ICU, assessed up to 30 days postoperatively.
  Intensive Care Unit (ICU) length of stay (LOS) is the duration (in days) a participant spends postoperatively in the ICU.
All-cause in-hospital 30-day mortality | From the date of surgery until death, assessed up to 30 days postoperatively.
  All-cause in-hospital 30-day mortality refers to death from any cause during the hospital stay within 30 days after cardiac surgery.
Postoperative pulmonary complications | Directly after cardiac surgery until the fifth postoperative day.
  Postoperative pulmonary complications (PPCs) are a composite of pulmonary events occurring within the first 5 postoperative days, including: - Mild respiratory failure: SpO₂ <90% or PaO₂ <7.9 kPa on room air, increased oxygen need, or oxygen use >2 days; - Severe respiratory failure: ventilatory support or hypoxemia despite oxygen; - Bronchospasm: new wheeze treated with bronchodilator; - Suspected infection: antibiotics plus new sputum, opacities, fever >38.3°C, or WBC >12,000/μL; - Pulmonary infiltrate: any unilateral or bilateral infiltrates on chest X-ray; - Aspiration pneumonitis: respiratory failure following inhalation of gastric contents; - Atelectasis: opacification with mediastinal shift and compensatory overinflation; - ARDS: as per global 2023 definition; - Pleural effusion: blunted costophrenic angle or hazy opacity; - Cardiopulmonary edema: congestion signs and interstitial infiltrates; and - Pneumothorax: air in pleural space with absent vascular markings.
Duration of mechanical ventilation | From the initiation of mechanical ventilation until the first discontinuation of mechanical ventilation, assessed up to 30 days postoperatively.
  Total duration (in hours) a patient peri-operatively receives support form a mechanical ventilator. Defined as the time (in hours) from intubation to the first extubation.

SECONDARY OUTCOMES:
Acute Kidney Injury (AKI) | Directly after cardiac surgery up to 30 days postoperatively.
  Incidence of Acute Kidney Injury as defined by the KDIGO 2012 criteria.
Postoperative stroke | Directly after cardiac surgery up to 30 days postoperatively.
  Post-operative stroke is defined as a cerebrovascular event (either ischemic or hemorrhagic) occurring within 30 days following cardiac surgery. The diagnosis is based on the onset of neurological deficits that may be temporary or persist long term, with confirmation via neuroimaging (CT or MRI) when possible.
Need for cardiac mechanical circulatory and/or cardiac, respiratory or cardiorespiratory extracorporeal life support modalities | Directly after cardiac surgery up to 30 days postoperatively.
  The incidence of postoperative use of cardiac mechanical circulatory (e.g. intra-aortic balloon pump, Impella) and/or cardiac, respiratory or cardiorespiratory extracorporeal life support (ECLS) modalities.
Postoperative Myocardial Infarction | Directly after cardiac surgery up to 30 days postoperatively.
  Postoperative myocardial infarction is a heart attack that occurs within the 30 days following cardiac surgery. The diagnosis requires evidence of new myocardial injury, primarily detected by an elevation in cardiac troponin or Creatine Kinase MB (CK-MB) levels, along with other clinical signs of ischemia like specific ECG changes or new wall motion abnormalities on imaging.
New-onset postoperative atrial fibrilliation | Directly after cardiac surgery up to 30 days postoperatively.
  New-onset postoperative atrial fibrillation is the development of atrial fibrillation within the first 30 days following cardiac surgery in participants who were not previously diagnosed with atrial fibrillation
Postoperative chest tube bloodloss | Measured in the first 12 hours after cardiac surgery
  Postoperative chest tube blood loss is the measured volume of blood drained from the chest cavity through surgically placed tubes following cardiac surgery.
Postoperative transfustion rates | Directly after cardiac surgery up to 30 days postoperatively.
  Defined as the number of units of erythrocytes (red blood cells), thrombocytes (platelets), and fresh frozen plasma (FFP) postoperatively transfused to each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Beukers, MD, PhD, Study Chair — Amsterdam UMC; David MP van Meenen, MD, PhD, Study Chair — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belway D, Tee R, Nathan HJ, Rubens FD, Boodhwani M. Temperature management and monitoring practices during adult cardiac surgery under cardiopulmonary bypass: results of a Canadian national survey. Perfusion. 2011 Sep;26(5):395-400. doi: 10.1177/0267659111409095. Epub 2011 May 18. PMID 21593083
- [Background] Klein A, Agarwal S, Cholley B, Fassl J, Griffin M, Kaakinen T, Mzallassi Z, Paulus P, Rex S, Siegemund M, van Saet A. A survey of patient blood management for patients undergoing cardiac surgery in nine European countries. J Clin Anesth. 2021 Sep;72:110311. doi: 10.1016/j.jclinane.2021.110311. Epub 2021 Apr 24. PMID 33905900
- [Background] Abbott TEF, Fowler AJ, Pelosi P, Gama de Abreu M, Moller AM, Canet J, Creagh-Brown B, Mythen M, Gin T, Lalu MM, Futier E, Grocott MP, Schultz MJ, Pearse RM; StEP-COMPAC Group. A systematic review and consensus definitions for standardised end-points in perioperative medicine: pulmonary complications. Br J Anaesth. 2018 May;120(5):1066-1079. doi: 10.1016/j.bja.2018.02.007. Epub 2018 Mar 27. PMID 29661384
- [Background] Authors/Task Force Members:; Jeppsson A; (Co-Chairperson) (Sweden); Rocca B; (Co-Chairperson) (Italy); Hansson EC; (Sweden); Gudbjartsson T; (Iceland); James S; (Sweden); Kaski JC; (United Kingdom); Landmesser U; (Germany); Landoni G; (Italy); Magro P; (Portugal); Pan E; (Finland); Ravn HB; (Denmark); Sandner S; (Austria); Sandoval E; (Spain); Uva MS; (Portugal); Milojevic M; (Serbia); EACTS Scientific Document Group. 2024 EACTS Guidelines on perioperative medication in adult cardiac surgery. Eur J Cardiothorac Surg. 2024 Dec 26;67(1):ezae355. doi: 10.1093/ejcts/ezae355. No abstract available. PMID 39385505
- [Background] Authors/Task Force Members; Kunst G, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Puis L, Wahba A; EACTS/EACTA/EBCP Committee Reviewers; Alston P, Fitzgerald D, Nikolic A, Onorati F, Rasmussen BS, Svenmarker S. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Br J Anaesth. 2019 Dec;123(6):713-757. doi: 10.1016/j.bja.2019.09.012. Epub 2019 Oct 2. No abstract available. PMID 31585674